CLINICAL TRIAL: NCT05625841
Title: Prevention and Improvement for Oral Mucositis Care During Chemoradiotherapy in Head and Neck Cancer Patients With Honey Production
Brief Title: Effects for Oral Mucositis Care During Chemoradiotherapy in Cancer Patients: Evaluation of the Bee Products
Acronym: Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: N2021100301
Record Dates: First submitted 2021-10-20; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Honey (Experimental): Each pack of 10 grams of honey after three meals a day.
  Interventions: Other: Honey product
- Honey and propolis (Experimental): Each pack contains 0.7ml of propolis + 9.3g of honey after three meals a day.
  Interventions: Other: Honey product; Other: propolis
- Usual care (Placebo Comparator): General routine oral care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Honey product — Bee products intervention from the first day of radiation to the end of radiation therapy duration 8-12 weeks.
  Arms: Honey; Honey and propolis
Other: propolis — propolis
  Arms: Honey and propolis
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
Oral mucositis is common among cancer patients receiving radiotherapy and chemotherapy. 80-90% of the patients are suffering from the mucositis pain; poor nutrition and even treatment discontinued. Some self-paid medications like glutamine has been used to prevent mucositis before and during radiotherapy/chemotherapy. Randomized controlled trials have shown that honey and propolis may be used for the management of mucositis. Honey demonstrates the most significant antibacterial effects; the green propolis has also been proved to comprise antibacterial, anti-inflammatory, and antioxidant effects. Bee products have been concerned as potential sources of natural antioxidants such as flavonoids, phenolic acids, and terpenoids. This study plan to conduct an RCT comparing the effectiveness of honey, honey and green propolis, and usual care in mucositis of cancer patients.

DETAILED DESCRIPTION:
Outcome Measures

1. Questionnaire collection: oral mucositis grade, pain scale, fatigue scale, dry mouth, nutritional status and quality of life scale.
2. Wearing the smart bracelet: The smart bracelet will automatically detect heart rate variability, heartbeat, sleep and activity status.
3. Saliva sample collection: Test the concentration of IL-1, IL-6, IL-10 and TNF in saliva.
4. Stool and oral flora collection: Test stool and oral flora microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with a head and neck tumor.
2. receive chemotherapy or radiotherapy.
3. conscious clear and willing to participate in the research.
4. can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

diabetes, arrhythmia, artificial heart rhythm device, allergic to bee products or alcohol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-11-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
oral mucositis severity | up to 12 weeks
  Ulceration or inflammation of the oral mucosa characterizes oral Mucositis

SECONDARY OUTCOMES:
pain score | up to 12 weeks
  visual analogue score(VAS)
fatigue level | up to 12 weeks
  Brief Fatigue Inventory
Xerostomia score | up to 12 weeks
  Xerostomia Inventory
nutrition level | up to 12 weeks
  Mini Nutritional Assessment
QoL questionnaire | up to 12 weeks
  FACT-HN
smart bracelet data | The first week, the fourth week, the 8th week start wearing the smart bracelet for 7 days
  The smart bracelet will automatically detect heart rate variability, heartbeat, sleep and activity status
Saliva specimen collection | This saliva is collected Baseline (before the start of radiotherapy), week 1, week 2, week 3, and up to 12 weeks
  Test the concentration of IL-1, IL-6, IL-10 and TNF in saliva
microbiota level | Baseline (Before the start of radiotherapy), week 2, week 4, and up to 12 weeks
  Stool and oral flora collection

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Wei Huang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No